CLINICAL TRIAL: NCT01837407
Title: Reconstruction of a Neurocutaneous Defect of the Proximal Phalanx With a Heterodigital Arterialized Nerve Pedicle Flap
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Tangshan (Other)
Collaborators: Chinese PLA General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: TSChen8871; HBTS13-04102 (Other: Ethics Committee of Hebei)
Record Dates: First submitted 2013-04-18; First posted 2013-04-23 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2011-06

CONDITIONS: Complex Digital Injuries
Keywords: Soft tissue loss; nerve defect; dorsal branch of the proper digital nerve; heterodigital arterialized nerve pedicle flap; Composite Flap; nerve flap; nerve transfer

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Surgical flap (Other): The flap includes the nerve for repair of the soft tissue and nerve defects
  Interventions: Procedure: Composite Flap

INTERVENTIONS:
Procedure: Composite Flap — nerve transfer with the dorsal branch of the digital nerve

SUMMARY:
Complex digital injuries involving soft tissue loss and digital nerve defect pose challenging problems for hand surgeons. This study uses the heterodigital arterialized nerve pedicle flap including the dorsal branch of the digital nerve for reconstructing a digital neurocutaneous defect of the proximal phalanx.

ELIGIBILITY:
Inclusion Criteria:

* a neurocutaneous defect at the proximal phalanx
* a soft tissue defect on the volar, dorsal, and contiguous lateral aspects of adjacent fingers .associated digital nerve defect.

Exclusion Criteria:

* an injury involving the course of the arterial or venous pedicle; an injury involving donor site or donor nerve
* a soft tissue defect on the noncontiguous lateral aspects of adjacent fingers
* a nerve injury that is able to be repaired by primary neurorrhaphy

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2008-03; Primary Completion 2011-09 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Static 2-point discrimination test | 18 months to 24 months
  The test points are at the center of the radial or ulnar portion of the pulp. Each area is tested 3 times with a Discriminator. The investigators stop at 4mm as a limit of 2PD and consider this normal.

SECONDARY OUTCOMES:
Cold Intolerance Severity Score (CISS) questionnaire. | 18 months to 24 months
  The maximum score is 100 and is grouped into 4 ranges (0-25, 26-50, 51-75, and 76-100), corresponding to mild, moderate, severe, and extreme severity, respectively.

OTHER OUTCOMES:
Visual analog scale | 18 months to 24 months
  The VAS consists of a 10-cm line that was grouped into mild (0-3 cm), moderate (4-6 cm), and severe (7-10 cm).

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Tangshan, Tangshan, Hebei, China

REFERENCES:
- [Result] Chen C, Zhang X, Shao X, Gao S, Wang B, Liu D. Treatment of a combination of volar soft tissue and proper digital nerve defects using the dorsal digital nerve island flap. J Hand Surg Am. 2010 Oct;35(10):1655-1662.e3. doi: 10.1016/j.jhsa.2010.07.011. PMID 20888502
- [Derived] Chen C, Tang P, Zhang X. Reconstruction of a neurocutaneous defect of the proximal phalanx with a heterodigital arterialised nerve pedicle flap. Injury. 2014 Apr;45(4):799-804. doi: 10.1016/j.injury.2013.09.034. Epub 2013 Sep 27. PMID 24125537